CLINICAL TRIAL: NCT00622362
Title: Depigmented and Polymerised Allergenic Extract of Dermatophagoides Pteronyssinus as Antiasthmatic Treatment for Children With Slight Allergic Asthma to Mites
Brief Title: Subcutaneous-Sublingual Immunotherapy With Depigmented and Polymerized Dermatophagoides Pteronyssinus Allergen Extract
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: Laboratorios Leti, S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2006-000571-15; 101-PG-COM-143
Record Dates: First submitted 2008-01-10; First posted 2008-02-25 (Estimated); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Allergic Asthma
Keywords: Immunotherapy; Allergy; Allergoid; Depigmented; Polymerized; Allergen-extract; mites; Asthma
MeSH Terms: conditions — Hypersensitivity; Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Active Comparator): Subcutaneous administration
  Interventions: Biological: DEPIGOID Dermatophagoides pteronyssinus
- B (Experimental): Sublingual administration
  Interventions: Biological: Polymerized TOL of Dermatophagoides pteronyssinus
- C (Placebo Comparator): Sublingual administration
  Interventions: Biological: Placebo Comparator

INTERVENTIONS:
Biological: DEPIGOID Dermatophagoides pteronyssinus — Subcutaneous administration:0.5 ml/month during 1 year
  Arms: A
Biological: Polymerized TOL of Dermatophagoides pteronyssinus — Sublingual immunotherapy. Two drops daily during 1 year
  Arms: B
Biological: Placebo Comparator — Sublingual immunotherapy. Two drops daily during 1 year
  Arms: C

SUMMARY:
The objective of this trial is to evaluate the clinical effectiveness of the administration of a depigmented and polymerized allergen extract Dermatophagoides pteronyssinus in children with allergic asthma due to this mite

DETAILED DESCRIPTION:
Immunotherapy is a specific treatment for allergic diseases. Unlike conventional pharmacological treatment, immunotherapy is the only treatment that could modify the natural course of allergic disease. This is a prospective double-blind placebo controlled study with three arms of treatment: placebo and two active (one of the active arms will receive subcutaneous immunotherapy and the other one will receive sublingual immunotherapy).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent signed by the patient and guardian.
* Positive clinical history of allergy to dust mites.
* FEV1 greater than or equal to 80% of the expected value and improvement in FEV1 greater than 12% after bronchodilation.
* Age-between 5 and 14 years.
* Sensitization to dust mites, diagnosed by positive skin tests to Dermatophagoides pteronyssinus: wheal size > 3 mm diameter and / or RAST (> 0.7 kU / L).

Exclusion Criteria:

* Patients out of the age range.
* Use of immunotherapy during the last four years.
* Any contraindication for the use of immunotherapy in accordance with European Allergy and Clinical Immunology Immunotherapy Subcommittee criteria:

  * Treatment with ß-blockers
  * Patients who have a condition in which adrenaline is contraindicated (hyperthyroidism, hypertension, heart disease, etc..).
  * Coexistence of immunopathological diseases (e.g. of the liver, kidney, the nervous system, thyroid gland, rheumatic diseases) in which autoimmune mechanisms play a role
  * Patients suffering from immune deficiencies
  * Patients with serious psychiatric / psychological disturbances
* Patients aspirin intolerance

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Symptom and medication scores | 1 year per patient

SECONDARY OUTCOMES:
Comparison between sublingual and subcutaneous administration route, quality of life, cost-effectiveness, dose response prick-test, inflammatory markers, exhaled nitric oxide, inflammatory markers in exhalate bronchial condensate, use of health resources | 1 year per patient
QoL | 1 year
  The Paediatric Asthma Quality of Life Questionnaire (PAQLQ) was developed to measure the functional problems (physical, emotional and social) that are most troublesome to children with asthmaQuestionnaire" E. Juniper
Cost-effectiveness | 1 year
Dose response prick-test | 1 year
Inflammatory markers | 1 year
Use of health resources | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Nieto, MD PhD, Principal Investigator
Locations (1):
- Hospital Universitario La Fé, Valencia, Spain